CLINICAL TRIAL: NCT01777061
Title: Clinical Management Decisions Based on [11C]Acetate Positron Emission Tomography Performed on Prostate Cancer Patients With Biochemical Recurrence
Brief Title: Clinical Management Decisions for Recurrent Prostate Cancer Patients Based on [11C]Acetate PET Scan
Status: No longer available | Type: Expanded Access
Sponsor: Wendell Yap, MD (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Sponsor-Investigator, Wendell Yap, MD, Assistant Professor, Department of Radiology, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 13429
Record Dates: First submitted 2013-01-17; First posted 2013-01-28 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Recurrent Prostate Cancer; PET Scan; FDG-PET; [11C]Acetate; C11-Acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — carbon-11 acetate; Sodium Acetate

INTERVENTIONS:
Drug: [11C]Acetate — intravenous injection of an average of 40 mCi of [11C]Acetate
  Other Names: carbon-11 acetate [[11C]acetate]; sodium acetate [11C]Acetate injection

SUMMARY:
When evaluating prostate cancer patients for recurrent disease, computed tomography (CT), and magnetic resonance imaging (MRI) are both highly sensitive methods for detecting lymph nodes, but are not specific as to whether the lymph nodes are malignant or benign.

While positron emission tomography (PET) utilizing radioactive glucose (FDG) has revolutionized staging, restaging, and monitoring response to therapy in many prevalent cancers such as breast, colorectal, esophageal, head and neck, lung, lymphoma, and melanoma, findings with prostate cancer have proven less sensitive because prostate cancer has a lower avidity for glucose. A newer PET isotope, utilizing acetate that is incorporated into the cell membrane of rapidly proliferating cells, has shown greater sensitivity than FDG in detecting prostate cancer.

This study will assess the clinical effectiveness of utilizing [11C]Acetate PET scans in identifying recurrent prostate cancer.

DETAILED DESCRIPTION:
FDG-PET imaging uses a form of radioactive glucose (18-fluoro-deoxyglucose or FDG), which allows the measurement of glucose metabolic rate of any tissue in the body. The most prevalent tumors have a glucose avidity that is typically greater than 2.5 times the avidity of benign tissue. Therefore, FDG-PET is able to discriminate between benign lymph nodes and those containing metastases, and similarly between scar tissue and recurrence of tumor.

Unfortunately, prostate cancer is only minimally glucose avid, and therefore, FDG-PET is much less effective in staging prostate cancer. The current FDA-approved imaging agent for prostate cancer is a monoclonal antibody specific for prostate cancer cells, capromab pendetide, labeled with a long-lived radionuclide [111]Indium that is used to image the patient over a six day period. However, recent data show that another PET radiopharmaceutical, [11C]Acetate (which has been FDA approved for years for cardiac imaging), is avidly taken up by prostate metastasis and is more sensitive than either [111]Indium capromab pendetide or FDG-PET.

This study will assess the clinical effectiveness of utilizing [11C]Acetate PET scans in identifying recurrent prostate cancer and aim to find at what PSA levels it is most effective.

ELIGIBILITY:
Inclusion Criteria:

* Positive for recurrent prostate cancer by PSA criteria
* Recurrence definition:
* Status post-operative radical prostatectomy, recurrence is defined by a PSA of greater than or equal to 0.2 ng/ml
* Patients who have failed external beam radiation, or status post-brachytherapy, have recurrence as defined as PSA above 2.0 ng/ml the nadir PSA after treatment
* Subject is able to comprehend the study objectives and provide written informed consent before the initiation of any study-related procedures.

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) status of ≥ 2
* Any other concurrent malignancy
* Patients without remission of disease (no PSA decrease)
* Patients without recurrence of disease (PSA remains low)

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Wendell Yap, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States